CLINICAL TRIAL: NCT04995640
Title: CILCA Registry: Aortic Arch Variant With a Common Origin of the Innominate and Left Carotid Artery. Management and Outcomes of Open and Endovascular Repair.
Brief Title: CILCA Arch Registry: Management and Outcomes of Open and Endovascular Repair
Status: Recruiting | Type: Observational
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Massimiliano M. Marrocco-Trischitta, Vascular surgeon, Ospedale San Donato
Other Study IDs: 163/int/2020
Record Dates: First submitted 2021-03-29; First posted 2021-08-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Aortic Arch; Aortic Diseases; Bovine Arch
Keywords: TEVAR; bovine arch; endovascular treatment; open surgery; aortic arch variant; aortic arch
MeSH Terms: conditions — Aortic Diseases | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CILCA patients: Subject with a CILCA and a thoracic cardiovascular disease requiring treatment. Both open cardiovascular repair and endovascular treatment (TEVAR) will be included.
  Interventions: Procedure: open cardiovascular repair or endovascular treatment (TEVAR)

INTERVENTIONS:
Procedure: open cardiovascular repair or endovascular treatment (TEVAR) — Surgery type: open cardiovascular repair and endovascular treatment (TEVAR)

SUMMARY:
This registry aims to provide insights on the pathogenic mechanisms that expose subjects with CILCA arch to the increased risk of postoperative complications. So, the CILCA arch registry will capture clinical data and medical images of subjects with CILCA arch treated by surgical or endovascular (TEVAR) means.

Study Design: International Multicenter and Observational registry

Estimated Enrolment: 500 patients, with competitive enrolment.

Clinical Follow up: Postoperatively at 30 days, at 12 months, and yearly after.

DETAILED DESCRIPTION:
The so-called "bovine" aortic arch (BAA) is characterized by the presence of a common origin of the innominate and left carotid artery, or, less frequently, by the origin of the left carotid directly from the innominate artery (i.e. type 2 BAA). In the present protocol, for brevity and according to the STROBE guidelines the investigators employed the acronym CILCA (common origin of the innominate and left carotid artery) arch, previously employed in publications of our group.

The CILCA is the second more common arch configuration, and its prevalence in the general population is 13.6%, with relevant differences among ethnic groups. However, the real prevalence of the CILCA is likely underestimated, because its presence is largely unreported due to the presumed clinical irrelevance of this anatomical variant. In fact, the peculiar anatomical features associated with the CILCA mandate specific management strategies and preoperative planning in both surgical and endovascular procedures involving the aortic arch, including type A aortic dissection repair and carotid stenting.

There is increasing evidence in the literature that the CILCA represents a potential determinant of the onset of thoracic aortic disease. Notably, it is associated with a 1.4-fold increased risk of developing aortic aneurysms or dissections, and this entails a relevant prevalence of this anatomical variant among patients requiring thoracic endovascular aortic repair (TEVAR). In fact, the CILCA presents a consistent and peculiar anatomical pattern compared with standard arch configuration, which provides relevant information for TEVAR planning, and may have prognostic implications.

This registry aims to provide insights on the pathogenic mechanisms that expose subjects with CILCA arch to the increased risk of postoperative complications. So, the CILCA arch registry will capture clinical data and medical images of subjects with CILCA arch treated by surgical or endovascular (TEVAR) means.

Technical and specific aims:

* Development of automatic segmentation of medical images for the assessment of geometric features by machine learning
* Assessment of a simplified method for the calculation of the "displacement forces" in proximal landing zones for TEVAR

Primary Endpoint: Identification of peculiar anatomical characteristics in patients with CILCA arch, before\after treatment of aortic pathologies (including both TEVAR and Open Repair).

Secondary Endpoint: Identification of anatomical risk factors for the postoperative clinical outcomes.

REGISTRY DESIGN International Multicenter and Observational clinical registry. Enrollment will include 500 patients with CILCA arch, treated with TEVAR or open repair. All patients will be followed up for 5 years, and their' clinical pathway and treatment strategy will be at discretion of the operator following current guidelines for thoracic aortic disease.

FOLLOW-UP PERIOD Postoperatively, patients will be followed-up for 5 years. This includes every medical check-up performed according to clinical practice (including telephone contacts) to obtain information regarding medical history, cardiovascular drugs use, hospitalizations, and adverse events, at 30 days, at 12 months, and yearly after. Repeated imaging (i.e. CT scan or magnetic resonance imaging) will be obtained according to current guidelines, or medical need.

STATISTICAL ANALYSIS All patients who are successfully registered will be included in the analysis. Being this an observational registry aiming to investigate the postoperative outcomes of patients with CILCA, the investigators proceeded without a formal power analysis. The number of patients scheduled to be enrolled (i.e. 500) was deemed adequate to provide robust evidence for future statistical analyses.

The study will be performed according to "good clinical practice ". The collection of personal, procedural and clinical data of patients must take place into the electronic CRF. Only the investigators and the personnel registered on the "Site Personnel Signature Log" will be granted access to the eCRF.

.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* CILCA arch treated for an aortic disease (i.e. aortic dissection, aneurysm)

Exclusion Criteria:

* Contraindications to computed tomography (e.g. hypersensitivity to contrast media, renal failure);
* Suspected or manifested pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with a CILCA and a thoracic cardiovascular disease requiring treatment. Both open cardiovascular repair and endovascular treatment (TEVAR) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Angulation of ascending aortic curvature | From Admission to 5 years follow-up
  Comparison among the Type of Arch (TOA), among pre- and post-Thoracic Endovascular Aortic Repair (TEVAR) or Open repair
Arch angle | From Admission to 5 years follow-up
  Comparison among the TOA, among pre- and post-TEVAR or Open repair
Centerline curvature radius (mm) | From Admission to 5 years follow-up
  Comparison among the TOA, among pre- and post-TEVAR or Open repair
Outer curvature radius (mm) | From Admission to 5 years follow-up
  Comparison among the TOA, among pre- and post-TEVAR or Open repair
Centerline tortuosity | From Admission to 5 years follow-up
  Comparison among the TOA, among pre- and post-TEVAR or Open repair
Volume of the ascending aorta (cm3) | From Admission to 5 years follow-up
  Comparison among the TOA, among pre- and post-TEVAR or Open repair

SECONDARY OUTCOMES:
Area of proximal landing zones (PLZs, mm2) | From Admission to 5 years follow-up
  Comparison among the TOA and PLZs; comparison among pre- and post-TEVAR or Open repair
Maximum diameter of PLZs (mm) | From Admission to 5 years follow-up
  Comparison among the TOA and PLZs; comparison among pre- and post-TEVAR or Open repair
Arch length of PLZs (mm) | From Admission to 5 years follow-up
  Comparison among the TOA and PLZs; comparison among pre- and post-TEVAR or Open repair
β angle of PLZs (°) | From Admission to 5 years follow-up
  Comparison among the TOA and PLZs; comparison among pre- and post-TEVAR or Open repair
Tortuosity angle (°) | From Admission to 5 years follow-up
  Comparison among the TOA and PLZs; comparison among pre- and post-TEVAR or Open repair

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Maria Marrocco-Trischitta, MD, PhD, Principal Investigator — Ospedale San Donato , IRCCS
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moorehead PA, Kim AH, Miller CP, Kashyap TV, Kendrick DE, Kashyap VS. Prevalence of Bovine Aortic Arch Configuration in Adult Patients with and without Thoracic Aortic Pathology. Ann Vasc Surg. 2016 Jan;30:132-7. doi: 10.1016/j.avsg.2015.05.008. Epub 2015 Jul 10. PMID 26166538
- [Background] Marrocco-Trischitta MM, Alaidroos M, Romarowski RM, Milani V, Ambrogi F, Secchi F, Glauber M, Nano G. Aortic arch variant with a common origin of the innominate and left carotid artery as a determinant of thoracic aortic disease: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2020 Mar 1;57(3):422-427. doi: 10.1093/ejcts/ezz277. PMID 31620770
- [Background] Rylski B, Pacini D, Beyersdorf F, Quintana E, Schachner T, Tsagakis K, Ronchey S, Durko A, De Paulis R, Siepe M, Roselli EE, Carrel T, Czerny M, Schoenhoff FS; EACTS Vascular Domain, EJCTS and ICVTS Editorial Committees. Standards of reporting in open and endovascular aortic surgery (STORAGE guidelines). Eur J Cardiothorac Surg. 2019 Jul 1;56(1):10-20. doi: 10.1093/ejcts/ezz145. PMID 31102528
- [Background] Marrocco-Trischitta MM, Romarowski RM, Alaidroos M, Sturla F, Glauber M, Nano G. Computational Fluid Dynamics Modeling of Proximal Landing Zones for Thoracic Endovascular Aortic Repair in the Bovine Arch Variant. Ann Vasc Surg. 2020 Nov;69:413-417. doi: 10.1016/j.avsg.2020.05.024. Epub 2020 May 29. PMID 32479874
- [Background] Marrocco-Trischitta MM, Alaidroos M, Romarowski RM, Secchi F, Righini P, Glauber M, Nano G. Geometric Pattern of Proximal Landing Zones for Thoracic Endovascular Aortic Repair in the Bovine Arch Variant. Eur J Vasc Endovasc Surg. 2020 May;59(5):808-816. doi: 10.1016/j.ejvs.2019.11.019. Epub 2019 Dec 27. PMID 31889656
- [Background] Popieluszko P, Henry BM, Sanna B, Hsieh WC, Saganiak K, Pekala PA, Walocha JA, Tomaszewski KA. A systematic review and meta-analysis of variations in branching patterns of the adult aortic arch. J Vasc Surg. 2018 Jul;68(1):298-306.e10. doi: 10.1016/j.jvs.2017.06.097. Epub 2017 Aug 31. PMID 28865978
- [Background] Hornick M, Moomiaie R, Mojibian H, Ziganshin B, Almuwaqqat Z, Lee ES, Rizzo JA, Tranquilli M, Elefteriades JA. 'Bovine' aortic arch - a marker for thoracic aortic disease. Cardiology. 2012;123(2):116-24. doi: 10.1159/000342071. Epub 2012 Sep 28. PMID 23037917
- [Background] Berko NS, Jain VR, Godelman A, Stein EG, Ghosh S, Haramati LB. Variants and anomalies of thoracic vasculature on computed tomographic angiography in adults. J Comput Assist Tomogr. 2009 Jul-Aug;33(4):523-8. doi: 10.1097/RCT.0b013e3181888343. PMID 19638843
- [Background] Maxwell BG, Harrington KB, Beygui RE, Oakes DA. Congenital anomalies of the aortic arch in acute type-a aortic dissection: implications for monitoring, perfusion strategy, and surgical repair. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):467-72. doi: 10.1053/j.jvca.2013.12.001. Epub 2014 Apr 14. PMID 24731741
- [Background] Faggioli GL, Ferri M, Freyrie A, Gargiulo M, Fratesi F, Rossi C, Manzoli L, Stella A. Aortic arch anomalies are associated with increased risk of neurological events in carotid stent procedures. Eur J Vasc Endovasc Surg. 2007 Apr;33(4):436-41. doi: 10.1016/j.ejvs.2006.11.026. Epub 2007 Jan 19. PMID 17240174
- [Background] Mylonas SN, Barkans A, Ante M, Wippermann J, Bockler D, Brunkwall JS. Prevalence of Bovine Aortic Arch Variant in Patients with Aortic Dissection and its Implications in the Outcome of Patients with Acute Type B Aortic Dissection. Eur J Vasc Endovasc Surg. 2018 Mar;55(3):385-391. doi: 10.1016/j.ejvs.2017.12.005. Epub 2018 Jan 12. PMID 29338980
- [Background] Shalhub S, Schafer M, Hatsukami TS, Sweet MP, Reynolds JJ, Bolster FA, Shin SH, Reece TB, Singh N, Starnes BW, Jazaeri O. Association of variant arch anatomy with type B aortic dissection and hemodynamic mechanisms. J Vasc Surg. 2018 Dec;68(6):1640-1648. doi: 10.1016/j.jvs.2018.03.409. Epub 2018 May 24. PMID 29804742
- [Background] Dumfarth J, Chou AS, Ziganshin BA, Bhandari R, Peterss S, Tranquilli M, Mojibian H, Fang H, Rizzo JA, Elefteriades JA. Atypical aortic arch branching variants: A novel marker for thoracic aortic disease. J Thorac Cardiovasc Surg. 2015 Jun;149(6):1586-92. doi: 10.1016/j.jtcvs.2015.02.019. Epub 2015 Feb 14. PMID 25802134
- [Background] Altnji HE, Bou-Said B, Walter-Le Berre H. Morphological and stent design risk factors to prevent migration phenomena for a thoracic aneurysm: a numerical analysis. Med Eng Phys. 2015 Jan;37(1):23-33. doi: 10.1016/j.medengphy.2014.09.017. Epub 2014 Oct 22. PMID 25456396
- [Background] Grabenwoger M, Alfonso F, Bachet J, Bonser R, Czerny M, Eggebrecht H, Evangelista A, Fattori R, Jakob H, Lonn L, Nienaber CA, Rocchi G, Rousseau H, Thompson M, Weigang E, Erbel R; European Association for Cardio-Thoracic Surgery (EACTS); European Society of Cardiology (ESC); European Association of Percutaneous Cardiovascular Interventions (EAPCI). Thoracic Endovascular Aortic Repair (TEVAR) for the treatment of aortic diseases: a position statement from the European Association for Cardio-Thoracic Surgery (EACTS) and the European Society of Cardiology (ESC), in collaboration with the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2012 Jul;42(1):17-24. doi: 10.1093/ejcts/ezs107. Epub 2012 May 4. No abstract available. PMID 22561652
- [Background] Chen CK, Liang IP, Chang HT, Chen WY, Chen IM, Wu MH, Sheu MH, Shih CC. Impact on outcomes by measuring tortuosity with reporting standards for thoracic endovascular aortic repair. J Vasc Surg. 2014 Oct;60(4):937-44. doi: 10.1016/j.jvs.2014.04.008. Epub 2014 May 10. PMID 24820894
- [Background] Ueda T, Takaoka H, Raman B, Rosenberg J, Rubin GD. Impact of quantitatively determined native thoracic aortic tortuosity on endoleak development after thoracic endovascular aortic repair. AJR Am J Roentgenol. 2011 Dec;197(6):W1140-6. doi: 10.2214/AJR.11.6819. PMID 22109332
- [Background] Marrocco-Trischitta MM, van Bakel TM, Romarowski RM, de Beaufort HW, Conti M, van Herwaarden JA, Moll FL, Auricchio F, Trimarchi S. The Modified Arch Landing Areas Nomenclature (MALAN) Improves Prediction of Stent Graft Displacement Forces: Proof of Concept by Computational Fluid Dynamics Modelling. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):584-592. doi: 10.1016/j.ejvs.2017.12.019. Epub 2018 Feb 6. PMID 29426592
- [Background] Marrocco-Trischitta MM, de Beaufort HW, Secchi F, van Bakel TM, Ranucci M, van Herwaarden JA, Moll FL, Trimarchi S. A geometric reappraisal of proximal landing zones for thoracic endovascular aortic repair according to aortic arch types. J Vasc Surg. 2017 Jun;65(6):1584-1590. doi: 10.1016/j.jvs.2016.10.113. Epub 2017 Feb 20. PMID 28222992
- [Background] Marrocco-Trischitta MM, Romarowski RM, de Beaufort HW, Conti M, Vitale R, Secchi F, Auricchio F, Trimarchi S. The Modified Arch Landing Areas Nomenclature identifies hostile zones for endograft deployment: a confirmatory biomechanical study in patients treated by thoracic endovascular aortic repairdagger. Eur J Cardiothorac Surg. 2019 May 1;55(5):990-997. doi: 10.1093/ejcts/ezy409. PMID 30535119